CLINICAL TRIAL: NCT00000696
Title: A Phase I/II Open Label Study To Evaluate the Antiviral Potential of Combination Low-Dose Therapy With Zidovudine and Interferon-Alpha 2A in Patients With Symptomatic HIV Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 068; 11042 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interferon Alfa-2a; Drug Therapy, Combination; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Interferon alpha-2; Zidovudine

INTERVENTIONS:
Drug: Interferon alfa-2a
Drug: Zidovudine

SUMMARY:
To evaluate the anti-HIV effect of single agent versus combination therapy with zidovudine (AZT) and interferon alfa-2a (IFN-A2a), as measured by p24 protein expression, viral growth and infectivity in patients with symptomatic HIV disease. To assess the safety of low dose schedules of AZT and IFN-A2a, alone and in combination, as measured by neutrophil counts and hepatic transaminase levels. To evaluate the comparative effects of single agent versus combination therapy with AZT and IFN-A2a on CD4 cell counts and skin test reactivity.

AZT is known to be an effective treatment for HIV infection. However, patients may develop reactions to AZT when it is administered for long periods of time. Combining AZT with another drug at lower doses might reduce toxicity in patients and prevent the development of drug resistant strains. IFN-A2a can reduce the growth of HIV in test tube experiments and recent studies have shown that when AZT and IFN-A2a are used together they reduce the growth of HIV more effectively than when either drug is used alone. This study will examine the effectiveness and safety of these drugs when they are given together and compare these results with the effectiveness and safety of the drugs when they are used alone.

DETAILED DESCRIPTION:
AZT is known to be an effective treatment for HIV infection. However, patients may develop reactions to AZT when it is administered for long periods of time. Combining AZT with another drug at lower doses might reduce toxicity in patients and prevent the development of drug resistant strains. IFN-A2a can reduce the growth of HIV in test tube experiments and recent studies have shown that when AZT and IFN-A2a are used together they reduce the growth of HIV more effectively than when either drug is used alone. This study will examine the effectiveness and safety of these drugs when they are given together and compare these results with the effectiveness and safety of the drugs when they are used alone.

AMENDED: 04-18-91 Treatment extended to 96 weeks. Patients are seen weekly for the first month and for the month following initiation of combination therapy (Cohorts 1, 2), then every other week until treatment week 48, followed by every week for the duration of the study. AMENDED: The doses have been modified to one of 4 total daily doses of AZT and one of 4 daily doses of IFN-A2a. AMENDED: Total treatment period will be 48 weeks. AMENDED: 9-24-90 Treatment will end 901214. Original Design: Before beginning any treatment, patients are carefully examined and evaluated. Each patient receives medication for 24 weeks, followed by a 4-week follow-up period. Patients are assigned randomly to one of four dosing schedules within one of three groups stratified according to whether or not they have ever received AZT and / or IFN-A2a:

* Group 1 receives AZT alone for 12 weeks, then AZT plus IFN-A2a for the following 12 weeks.
* Group 2 receives IFN-A2a alone for 12 weeks, then IFN-A2a plus AZT for the following 12 weeks.
* Group 3 receives the combination of AZT and IFN-A2a for 24 weeks. Medications are administered according to one of four possible daily dosing schedules of AZT plus IFN-A2a (increasing doses of each). AZT is taken by mouth as a capsule every 6 hours. IFN-A2a is given by an injection under the skin once a day. Initially, doses of IFN-A2a are given by one of the research staff, after which patients are taught to give their own injections. Patients are examined weekly for the first 4 weeks, then every other week until the end of the study. Patients assigned to groups receiving two drugs will be examined weekly again for 4 weeks when the second drug is added.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP), as aerosolized pentamidine.
* Ibuprofen.
* Acute therapy (7 days) with oral acyclovir.
* Acute therapy with ketoconazole.

Patients must have:

* A diagnosis of AIDS related complex as well as defined symptoms within 12 months of study entry in the absence of concurrent illness or conditions other than HIV infection.
* Estimated life expectancy of at least 12 weeks.
* Positive serum p24 antigen > 70 pg/ml. Patients may have received prior zidovudine (AZT) and / or interferon alpha therapy, provided that:
* The total duration of treatment was < 6 months. Patients treated > 12 weeks but < 6 months should have received continuous therapy (no more than 14 consecutive days or 21 total days off during the treatment period). For patients treated = or < 12 weeks, continuous treatment means < 7 days off total during the treatment period. For all patients, a washout period of = or > 4 weeks must have elapsed prior to study entry. Treatment did not result in a major adverse reaction attributable to AZT or IFN-A2a such that rechallenge at a randomly assigned dosage level would be precluded.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Acquired immunodeficiency syndrome (AIDS) as defined by opportunistic infections.
* Significant cardiac (New York Heart Association Class 3 or 4), hepatic, renal, or neurologic disorder.
* Concurrent neoplasm other than basal cell carcinoma or in situ carcinoma of the cervix.
* Significant neurological disorder which impairs the patient's ability to give or receive informed consent or reduces the patient's performance status to the extent that protocol requirements and self-administration of drug cannot be accurately completed.

Concurrent Medication:

Excluded:

* All concomitant medications should be kept to a minimum.
* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP), other than aerosolized pentamidine.
* Other antiretroviral agents.
* Experimental medications.
* Biologic response modifiers.
* Systemic corticosteroids.
* Cimetidine.
* Ranitidine.
* Aspirin, acetaminophen, and nonsteroidal anti-inflammatory agents with the exception of ibuprofen.
* Barbiturates.
* Cardiac glycosides, antiarrhythmics, or vasodilators.
* Systemic treatment for an active infection, including pulmonary tuberculosis.

Concurrent Treatment:

Excluded:

* Systemic treatment for an active infection, including pulmonary tuberculosis.

Patients with the following will be excluded from the study:

* AIDS as defined by opportunistic infections, Kaposi's sarcoma, or other AIDS defining neoplasms, HIV dementia complex, or HIV wasting disease.
* HIV constitutional disease. Any one of the following:
* Fever of > 38.5 degrees persisting for > 1 month.
* Involuntary weight loss of = or > 10 lbs or 10 percent of body weight.
* Diarrhea defined as = or > 2 liquid stools per day persisting for at least a total of 14 days without definable cause.
* Significant cardiac (New York Heart Association Class 3 or 4), hepatic, renal, or neurologic disorder.
* Concurrent neoplasm other than basal cell carcinoma or in situ carcinoma of the cervix.
* Significant neurological disorder which impairs the patient's ability to give or receive informed consent or reduces the patient's performance status to the extent that protocol requirements and self-administration of drug cannot be accurately completed.
* Prior AZT or IFN-A2a therapy for = or > 6 months.
* Previous major adverse reaction to AZT or IFN-A2a.

Prior Medication:

Excluded:

* Prior zidovudine (AZT) or interferon therapy for = or > 6 months.
* Excluded within 4 weeks of study entry:
* Any antiretroviral agent, Cytotoxic chemotherapy, or immunomodulator, including corticosteroids.
* Excluded within 30 days of study entry:
* Anti-infectives or agents likely to produce hematologic side effects (e.g., trimethoprim / sulfamethoxazole).
* Excluded: Cardiac glycosides, antiarrhythmics, or vasodilators.

Active substance abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Study Completion 1993-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D Mildvan, Study Chair
Locations (6):
- United States (6):
  - USC CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York

REFERENCES:
- [Background] Zucker ML, Huberman KT, Hirschman SZ, Mildvan D. Stability of HIV-1 p24 antigen upon prolonged storage at -70 degrees C. The ACTG 068 Collaborative Team. Int Conf AIDS. 1992 Jul 19-24;8(3):44 (abstract no PuA 6203)
- [Background] Mildvan D, Bassiakos Y. Zidovudine (ZDV) and interferon-alpha 2a (IFN): ongoing assessment of synergy and tolerance in early ARC patients, ACTG 068. The ACTG 068 Collaborative Group. Int Conf AIDS. 1992 Jul 19-24;8(2):B184 (abstract no PoB 3586)
- [Background] Mildvan D, Ruprecht R, Krown S, Pettinelli C. Methodological issues in AIDS clinical trials. Application of the combination index method in the design of a clinical antiretroviral trial: ACTG 068. J Acquir Immune Defic Syndr (1988). 1990;3 Suppl 2:S111-3 discussion S114-9. No abstract available. PMID 2231291
- [Background] Mildvan D, Bassiakos Y, Zucker ML, Hyslop N Jr, Krown SE, Sacks HS, Zachary J, Paredes J, Fessel WJ, Rhame F, Kramer F, Fischl MA, Poiesz B, Wood K, Ruprecht RM, Kim J, Grossberg SE, Kasdan P, Berge P, Marshak A, Pettinelli C. Synergy, activity and tolerability of zidovudine and interferon-alpha in patients with symptomatic HIV-1 infection: AIDS Clincal Trial Group 068. Antivir Ther. 1996 Apr;1(2):77-88. PMID 11321183